CLINICAL TRIAL: NCT06110117
Title: Open Clinical Investigation to Evaluate Efficacy and Safety of the Medical Device "Sterimar Stop & Protect Irritation & Dryness" in Adults With Dry or Irritated Nose
Brief Title: Assess Efficacy and Safety of a Nasal Spray in Adults With Dry or Irritated Nose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Church & Dwight Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST-22-U62
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-02

CONDITIONS: Dry Nose
MeSH Terms: interventions — Desiccation

STUDY DESIGN:
Intervention Model Description: Subjects will be evaluated for symptom severity before and during use of the nasal spray product.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nasal Spray (Experimental): 1 to 2 sprays per nostril of Sterimar Stop & Protect Irritation & Dryness for a minimum of 2 times (morning and evening) and, as needed, up to a maximum of 6 times per day (i.e. maximum 12 sprays per nostril each day) for seven days.
  Interventions: Device: Sterimar Stop & Protect Irritation & Dryness

INTERVENTIONS:
Device: Sterimar Stop & Protect Irritation & Dryness — One or two nasal sprays will be administered to each nostril for a minimum of 2 times per day up to a maximum of 6 times per day for seven days.

SUMMARY:
The goal of this clinical trial is to test symptom relief in subjects suffering from irritated or dry nasal passages. The main question it aims to answer is whether use of the nasal spray provides relief from dry nose symptoms. Participants will use the product for one week and report on the severity of their symptoms before and during use.

DETAILED DESCRIPTION:
The aim of this clinical investigation is to evaluate the efficacy and safety of a product among subjects suffering from the irritated or dry nasal mucosa triggered by any causes. Sterimar Stop & Protect Irritation & Dryness, similar to other nasal saline solutions, can clean the nose and eliminates impurities, restores natural moisture, and helps prevent ear, nose, and throat (ENT) disorders, consequently improving the quality of life. The test product is a seawater-based nasal spray enriched with sodium thiosulfate pentahydrate and sodium hyaluronate and is currently marketed in France. The current study is to evaluate the clinical benefits associated with using Sterimar Stop & Protect Irritation & Dryness in the relief of nasal dryness and irritation symptoms triggered by any causes.

60 subjects will be included in this single arm open label study.

Study product will be used as 1 to 2 sprays per nostril (each "dose" is 1 or 2 sprays per nostril, the second spray only if needed), for a minimum of 2 times (morning and evening) and, as needed, up to a maximum of 6 times per day (i.e., maximum 12 sprays per nostril each day) for seven days.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects ≥18 years of age;
2. Subjects must have ongoing nasal irritation or dryness at Visit 1 (Day -4);
3. Total Irritation Score (sum of all 12 symptom scores) must average at least 8 over the three-day run-in period (Day -3 to -1) and must be at least 8 at Visit 2 (Day 0). (Individual symptom score range is 0 - 3; Total Irritation Score range is 0 - 36.)
4. Dry Nose Symptom Score must average at least 2 over the three-day run-in period and must be at least 2 at Visit 2 (Day 0). (Dry nose symptom score range is 0 - 3.)
5. The score of at least two other symptoms beside dry nose must average at least 2 over the three-day run-in period and must be at least 2 at Visit 2 (Day 0). (Each symptom score range is 0 - 3.)
6. Twenty-five percent of the included subjects must have ongoing nasal symptoms caused by indoor pollutants from fireplaces, candles, smoking, or cooking, verified by principal investigator;
7. Subjects are willing to refrain from using any medications and/or acts for relief of nasal symptoms during the whole study from Day -4 to Day 7; except for acetaminophen, ibuprofen, or vitamins;
8. Subjects are willing and able to comply with the requirements of the study to use the study product according to use instructions, complete the daily symptom and product diaries and questionnaire(s), and visit the test facility as instructed;
9. Subjects can read, understand, and sign an informed consent document after being advised of the nature of the study.

Exclusion Criteria:

1. Currently taking any over-the-counter and prescription systemic/topical corticosteroids, antibiotics, antihistamines, cromone, nonsteroidal anti-inflammatory drugs (NSAIDs), leukotriene antagonists or topical or systemic decongestants within the two weeks prior to Visit 1;
2. Currently using other nasal sprays, nasal pumps, nasal irrigation/lavage devices, or oils, creams, or gels into the nose;
3. Women who are pregnant and/or breastfeeding or planning to become pregnant during the study and within 30 days after the last application of the study product;
4. Have a dermatologic, respiratory, or medical condition (e.g., asthma, pneumonia, laryngotracheobronchitis, sinusitis, etc.) which, in the opinion of the principal investigator, could interfere with the interpretation of study results at the time of the screening visit (Day -4);
5. Have a positive medical history of any significant illness within the 2 weeks prior to the screening visit (Day -4), which, in the opinion of the principal investigator, could interfere with the interpretation of study results;
6. Have a known allergy to any food or personal care products;
7. Have any kind of immunodeficiency;
8. Have a history of sensitivity to products as related to the product being evaluated;
9. Positive Coronavirus disease (COVID-19) test during the month before the study or during the study;
10. Self-reported history of anaphylaxis;
11. Confirmed diagnosis of urticaria or eczema;
12. Confirmed diagnosis of asthma that requires more than intermittent rescue beta-agonist treatment, for example, before exercise;
13. Immunotherapy during the past two years or ongoing immunotherapy;
14. Recent nasal or sinus surgery within the last six months;
15. Use of other nasal spray, pump, continuous positive airway pressure machine, nasal irrigation/lavage device, internal nasal gel, or nasal oil within 2 weeks before the screening visit (Day -4);
16. Presence of nasal polyposis and chronic sinusitis (assessed by the PI);
17. Nasal anatomic abnormality, e.g., severely deviated septum, congenital cleft lip/palate, nasal bleeding diathesis (assessed by the PI); and/or
18. Any clinically significant co-morbid condition, which, in PI's opinion, may affect the subject's safety and/or participation in the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-11-04 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported total irritation score from baseline | One week of product use.
  Sum of scores of 12 symptoms: nasal dryness, nasal crusting, nasal bleeding, nasal itching, nasal burning, nasal obstruction, nasal pain, nasal discomfort, sneezing, reduced sense of smell, external nasal redness, and external nasal swelling. Total score ranges from 0 to 36 in 0.5 unit increments with higher scores indicating more severe symptoms. (Lower is better)

SECONDARY OUTCOMES:
Change in patient-reported symptom score from baseline for each of the 12 symptoms from baseline to day 7. | One week of product use.
  7-point scale from 0 to 3 in 0.5-unit increments with higher scores indicating more severe symptoms. (Lower is better) nasal dryness, nasal crusting, nasal bleeding, nasal itching, nasal burning, nasal congestion, nasal pain, nasal discomfort, sneezing, reduced sense of smell, external nasal redness, external nasal swelling
Change in patient-reported quality of life question from baseline to day 7. | One week of product use.
  5-point scale for seven questions, plus one yes/no question. Scores range from 1 (very good) to 5 (very poor) in 1 unit increments. Yes/no on whether symptoms would have been treated if not in the study (yes means symptoms severe enough to treat).
Day on which a state of well-being of nose was achieved. | One week of product use.
  Day 0 to Day 7 or not at all.
Change from baseline in morning/evening total irritation and individual symptom scores. | One week of product use.
  Each symptom on a 7-point scale from 0 to 3 in 0.5-unit increments with higher scores indicating more severe symptoms. (Lower is better) Sum of symptom scores is total irritation score.
Immediate relief for individual symptom scores after first product application of the day. | 1 minute, 10 minutes, and 1 hour after first application on day 0 and on day 6.
  Each symptom on a 7-point scale from 0 to 3 in 0.5-unit increments with higher scores indicating more severe symptoms. (Lower is better)
Duration of relief of first dose each day. | One week of product use.
  Time between first and second product application of the day.
Change from baseline in sleep disturbance scores | One week of product use.
  Assessment of quality of sleep will be evaluated by means of a questionnaire ("Quality of Sleep Questionnaire"), on a 0 to 3-point scale, with higher score indicating a worse outcome, with 0=not at all, 1=slightly, 2=moderately and 3=severely, to be completed from Day 0 (baseline) and daily from the beginning to the end of the study.
Change from baseline in examiner symptom scores for dryness, atrophy, redness, oedema, crusting, and bleeding. | One week of product use.
  Each symptom on a 7-point scale from 0 to 3 in 0.5-unit increments with higher scores indicating more severe symptoms. (Lower is better)

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Eurofins Dermscan Poland, Gdansk
  - Centrum medyczne, Sztum

IPD SHARING:
Plan to Share IPD: No